CLINICAL TRIAL: NCT02234635
Title: Phase 1 Evaluate the Visual Quality Change of Eyes Implanted With Multifocal Intraocular Lens and Monofocal Lenses; Phase 2 Evaluate the Tear Film Quality Dynamics of Eyes Implanted With Multifocal Intraocular Lens and Monofocal Lenses.
Brief Title: Visual Quality Change of Eyes Implanted With Diffractive Multifocal Intraocular Lens After Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, yin ying zhao, doctor of ophthalmology, Principal Investigator, Clinical Professor, Wenzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VQIOL-21
Record Dates: First submitted 2014-07-31; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Dry Eye; Vision Disorders; Quality of Life
Keywords: visual acuity; objective visual quality; multifocal intraocular lens; tear-film quality dynamics
MeSH Terms: conditions — Dry Eye Syndromes; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- monofocal IOLs group (Other): monofocal IOLs group were implantation with Tecnis® ZCB00
  Interventions: Other: Diffractive multifocal IOLs group
- Diffractive multifocal IOLs group (Active Comparator): Diffractive multifocal IOLs group were implantation with Tecnis® ZMB00
  Interventions: Other: Diffractive multifocal IOLs group

INTERVENTIONS:
Other: Diffractive multifocal IOLs group — Diffractive IOLs are a type of multifocal (bifocal) IOL that are based on the Huygens-Fresnel principle. Specifically, a diffractive IOL has concentric rings in its posterior surface that form 2 primary focal points independent of pupil size. This optical behavior of the IOL can effectively restore far and near vision. However, it can also cause side effects, such as halos and glare and loss of contrast sensitivity.

SUMMARY:
In this study, the investigators examined the subjective visual quality including LogMAR uncorrected distance visual acuity (UCDVA), best corrected distance visual acuity (BCDVA),uncorrected intermediate visual acuity (UCIVA), distance corrected intermediate visual acuity (DCIVA), uncorrected near visual acuity (UCNVA) ,distance corrected near visual acuity (DCNVA),using logMAR visual acuity chart,and the objective visual quality including Modulation Transfer Function (MTF), Strehl ratio(SR), objective scatter index (OSI), OQAS value (OV),and the tear-film quality dynamics including the tear break-up time and the tear-film OSI between the eyes with multifocal lens and monofocal lenses by optical quality analysis system (OQAS).

DETAILED DESCRIPTION:
50 eyes of 50 cataract patients scheduled for phacoemulsification surgery were recruited, the multifocal group (25 eyes) ，were implantation with Tecnis® ZMB00；and the monofocal group (25 eyes) were implantation with Tecnis® ZCB00.

Methods: All eyes were examined by logMAR visual acuity chart and Optical quality analysis system (OQAS) at 1 week, 1 month, 3 month, 6 month,12 month after surgery for the subjective and objective visual quality Change during the first year.

Measures:Subjective and objective visual quality were evaluated.Tear-film quality dynamicswere evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with an axial length of 22.00 to 25.00 mm with age-related cataract.

Exclusion Criteria:

* Preoperative exclusion criteria included diabetes, history of ocular surgery or inflammation.
* Patients who could not be available for follow-up.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-09 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the Visual Quality Change of Eyes Implanted With Diffractive Multifocal Intraocular Lens | 1week, 1month, 3month,6month,12month
  Visual quality change during the first year after cataract surgery. The visual quality including the subjective and objective visual quality. The subjective visual quality including LogMAR uncorrected distance visual acuity (UCDVA), best corrected distance visual acuity (BCDVA),uncorrected intermediate visual acuity (UCIVA), distance corrected intermediate visual acuity (DCIVA), uncorrected near visual acuity (UCNVA) and distance corrected near visual acuity (DCNVA).
  The objective visual quality including Modulation Transfer Function (MTF), Strehl ratio(SR), objective scatter index (OSI) and OQAS value (OV).

SECONDARY OUTCOMES:
To evaluate the Tear-film Quality Dynamics of Eyes Implanted With Diffractive Multifocal Intraocular Lens | 1week, 1month, 3month,6month,12month
  The tear-film quality dynamics including the tear break-up time and the tear-film OSI were examined by optical quality analysis system (OQAS)

CONTACTS AND LOCATIONS:
Overall Officials: Fang Yu, Study Director — Affiliated Eye Hospital of Wenzhou Medical University
Locations (1):
- Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Ye L, Chen T, Hu Z, Yang Q, Su Q, Li J. Comparison of the visual performance between Oculentis MF30 and Tecnis ZMB00 multifocal intraocular lenses. Ann Transl Med. 2021 Jan;9(2):144. doi: 10.21037/atm-20-7777. PMID 33569446
- [Derived] Chen T, Yu F, Lin H, Zhao Y, Chang P, Lin L, Chen Q, Zheng Q, Zhao YE, Lu F, Li J. Objective and subjective visual quality after implantation of all optic zone diffractive multifocal intraocular lenses: a prospective, case-control observational study. Br J Ophthalmol. 2016 Nov;100(11):1530-1535. doi: 10.1136/bjophthalmol-2015-307135. Epub 2016 Feb 22. PMID 26903522